CLINICAL TRIAL: NCT06593457
Title: A Phase 1, 2-Part, Placebo-Controlled, Double-Blinded Study to Assess the Effect of Food and Drug-Drug Interaction of Fluconazole on the Pharmacokinetics of NX-5948
Brief Title: A Food-Effect, Drug-Drug Interaction, and Pharmacokinetics Study of NX-5948 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NX-5948-302
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: Drug-Drug Interaction; Food effects; Healthy participants; Pharmacokinetics; Pharmacodynamics; NX-5948; BTK Degrader

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Sequence 1 (Treatment A, B, C) (Experimental): Period 1: NX-5948 or placebo administered under fasted conditions Period 2: NX-5948 or placebo administered under fed conditions Period 3: Fluconazole and single dose of NX-5948/placebo coadministered on Day 4
  Interventions: Drug: IP; Drug: Matching Placebo
- Part 1: Sequence 2 (Treatment B, A, C) (Experimental): Period 1: NX-5948 or placebo administered under fed conditions Period 2: NX-5948 or placebo administered under fasted conditions Period 3: Fluconazole and single dose of NX-5948/placebo coadministered on Day 4
  Interventions: Drug: IP; Drug: Matching Placebo
- Part 2: NX-5948 PK (Experimental): Experimental: Part 2: NX-5948 PK NX-5948 or placebo administered 2 doses given 12 hours apart under fasted conditions
  Interventions: Drug: IP; Drug: Matching Placebo

INTERVENTIONS:
Drug: IP — NX-5948 oral
Drug: Matching Placebo — Fluconazole

SUMMARY:
This is a Phase 1, 2-part double-blinded (with respect to NX-5948/placebo), placebo-controlled study. Part 1 is a randomized, 3 period cross-over food-effect (FE) and drug-drug interaction (DDI) study. Part 2 is a single-period PK evaluation study.

DETAILED DESCRIPTION:
Part 1:

Periods 1 and 2: Subjects will be randomized to 1 of 2 treatment sequences in a 1:1 ratio. In each treatment sequence, subjects will be randomized to receive either active NX-5948 or placebo in a 7:2 ratio. Subjects will receive a single dose of NX-5948 or placebo under fasting or fed conditions as per randomization schedule to evaluate the effect of food on the single- dose pharmacokinetics (PK) of NX-5948 in healthy subjects.

Period 3: Fluconazole will be administered every day for 8 consecutive days with a single dose of NX-5948/placebo coadministered on Day 4 to evaluate the effect of fluconazole on the single dose PK of NX-5948 in healthy subjects.

Part 2:

Subjects will be randomized to receive either active NX-5948 or placebo to assess single-period PK.

Parts 1 and 2: Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

* Healthy, adult, male, 18-55 years of age
* Subjects must follow protocol-specified contraception guidance as described in the protocol.
* Continuous non-smoker who has not used nicotine and tobacco containing products for at least 3 months prior to the first dosing based on subject self-reporting.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and 12-lead safety ECGs, at the screening visit and/or first check-in, as deemed by the PI or designee,
* Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

Key Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any of the following criteria:

* Clinically significant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neoplastic (including leukemia, lymphoma, malignant melanoma), myeloproliferative, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine or connective tissue diseases or disorders, or any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the subjects by their participation in the study.
* History or presence of hypersensitivity, angioedema, or idiosyncratic reaction to the study drug(s) or related compounds.
* History or presence of:

  * Significant multiple and/or severe allergies, including anaphylactic reaction.
  * Risk factors for Torsade de Pointes (e.g., heart failure, cardiomyopathy, family history of Long QT Syndrome, or sudden unexpected cardiac death at a young age).
  * Sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities.
  * Myocardial infarction, acute coronary syndrome, cerebrovascular accident, transient ischemic attack, clinically significant ventricular or atrial tachyarrhythmia as determined by the PI or designee, documented syncope without identified and corrected cause, a pacemaker or implantable cardioverter-defibrillator, cardiac or carotid/cerebral stent placement or angioplasty, or clinically significant valvular heart disease.
  * Adrenal insufficiency.
  * Skin infection.
* Positive Coronavirus disease 2019 (COVID-19) results at first check-in.
* Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit.
* Unable to refrain from or anticipates the use of:

  * Any drugs, including prescription and non prescription medications, herbal remedies, or vitamin supplements (including kava, ginko biloba, yohimbe, and saw palmetto) beginning 14 days prior to the first dosing.
  * Any drugs known to be moderate or strong inducers and inhibitors of CYP3A4, P gp, and/or breast cancer resistance protein, including St. John's Wort, dehydroepiandrosterone, and ginseng, beginning 28 days prior to the first dosing.
  * Any acid reducing agents beginning 7 days prior to the first dosing.
* Participation in another clinical study within 30 days or within 5 half-lives (if known), prior to the first dosing, whichever is longer. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients must be assigned the male gender at birth.
Enrollment: 32 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Part 1 Food Effect: AUC0-t for NX-5948 administered under fed and fasted conditions | 9 weeks
  To evaluate the effect of food on the single-dose pharmacokinetics (PK) of NX-5948 in healthy subjects.
Part 1 Food Effect: AUC0-inf for NX-5948 administered under fed and fasted conditions | Approximately 9 weeks
  To evaluate the effect of food on the single-dose pharmacokinetics (PK) of NX-5948 in healthy subjects.
Part 1 Food Effect: Cmax for NX-5948 administered under fed and fasted conditions | 9 weeks
  To evaluate the effect of fluconazole on the single dose PK of NX-5948 in healthy subjects.
Part 1 Drug Drug Interaction: AUC0-inf for NX-5948 administered with and without fluconazole | 9 weeks
  To evaluate the effect of fluconazole on the single dose PK of NX-5948 in healthy subjects.
Part 1 Drug Drug Interaction: Cmax for NX-5948 administered with and without fluconazole | 9 weeks
  To evaluate the effect of fluconazole on the single dose PK of NX-5948 in healthy subjects.
Part 1 Drug Drug Interaction: AUC0-t for NX-5948 administered with and without fluconazole | Approximately 9 weeks
  To evaluate the effect of fluconazole on the single dose PK of NX-5948 in healthy subjects.
Part 2 PK: AUC0-inf for NX-5948 administration | 6 weeks
  To evaluate the PK of NX-5948 following 2 doses of NX-5948 given 12 hours apart in healthy subjects.
Part 2 PK: Cmax for NX-5948 administration | 6 weeks
  To evaluate the PK of NX-5948 following 2 doses of NX-5948 given 12 hours apart in healthy subjects.
Part 2 PK: AUC0-t for NX-5948 administration | Approximately 6 weeks
  To evaluate the PK of NX-5948 following 2 doses of NX-5948 given 12 hours apart in healthy subjects.

SECONDARY OUTCOMES:
Part 1: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Approximately 9 weeks
  To evaluate safety and tolerability of single doses of NX-5948 administered alone under fed and fasting conditions and following multiple doses of fluconazole in healthy subjects.
Part 2: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Approximately 6 weeks
  To evaluate safety and tolerability of 2 doses of NX-5948 given 12 hours apart in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Injac, MD PhD, Study Director — Nurix Therapeutics, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No